CLINICAL TRIAL: NCT03128307
Title: In-Home Study of Intraoral Device for Reducing Snoring Among Habitual Snorers
Brief Title: OTC Mouthpiece for Snoring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zyppah, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Zyppah01
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Intervention Model Description: Patient serves as their own control
Who Masked: Care Provider, Investigator
Masking Description: The data is compiled and analyzed by an outside, independent organization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Zyppah Anti-snoring Appliance — Use of an OTC mouth guard at night to prevent snoring

SUMMARY:
Online patient registration to participate in clinical trial to test OTC mouthpiece that controls position of the tongue to reduce snoring.

DETAILED DESCRIPTION:
Patient will complete informed consent, inclusion/exclusion criteria, sleep apnea and snoring surveys online. If patient meets all criteria for the study, patient will be provided with a treatment device for use for a 10 day treatment period. Patient will complete the trial upon providing final online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Living in the United States
* Signing the Informed Consent Form

Exclusion Criteria:

* Missing teeth (as the device won't be properly fitted)
* Any severe breathing or respiratory disorder, such as chronic asthma, emphysema, COPD, or a similar condition
* Poor dental health, such as severe gum disease, loose teeth, an abscess, mouth sores, or bleeding gums
* A dental implant placed within the last three months
* Diagnosed with a Temporomandibular joint condition (TMJ)
* Actively experiencing any mouth or jaw pain, including clenching of the teeth, grinding, or any other physical injury to the jaw or teeth
* Full dentures
* Braces
* Diagnosis of sleep apnea
* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Greenburg, DDS, Principal Investigator — Zyppah, Inc.
Locations (1):
- The EyeDeas Company, Lake Forest, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited online. A total of 764 expressed interest in the trial. 143 potential subjects either opted not to participate or did not meet the inclusion/exclusion criteria.
Groups:
- Clinical Trial Participants: Subjects who received the Zyppah Anti-Snoring device and were entered into the clinical study. Subjects were asked to use the device for ten consecutive nights and then fill out an online form assessing their experience with the device.
Period: Overall Study
Arm/Group | Clinical Trial Participants
Started | 604
Completed | 570
Not Completed | 34
Not completed — Lost to Follow-up | 29
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Clinical Trial Participants
Number analyzed (Participants) | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 465
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Snoring Severity Scale (1-9) [Mean (Standard Deviation); unit: units on a scale] — The Snoring Severity Scale (SSS) is a 9-point, validated scale to measure the severity of snoring. A total of three questions are asked: 1) "How often do you snore, 2) "How long do you snore", and 3) How audible is your snoring. Answers for each of these questions are summed for a total SSS score. A score of '0' would indicate no snoring at all, while a score of '9' would indicate the most severe snoring as measured by the SSS.
  units on a scale | 6.2 (1.57)
How Much Does your Snoring bother YOU: VAS (1-10) [Mean (Standard Deviation); unit: units on a scale] — A visual-analogue scale (VAS) was used to measure how much snoring bothered the individual user. A score of '0' was not bothersome at all, while a score of '10' would indicate it is extremely bothersome.
  units on a scale | 5.08 (2.91)
How Much Does your Snoring bother YOUR PARTNER: VAS (1-10) [Mean (Standard Deviation); unit: units on a scale] — A visual-analogue scale (VAS) was used to measure how much snoring bothered the subject's partner (if applicable). A score of '0' was not bothersome at all, while a score of '10' would indicate it is extremely bothersome.
  units on a scale | 8.92 (1.98)
How Frequently Do you Snore: VAS (1-10) [Mean (Standard Deviation); unit: units on a scale] — A visual-analogue scale (VAS) was used to measure how frequently the subject snored. A score of '0' would indicate the subject never snored, while a score of '10' would indicate the subject snores every single night.
  units on a scale | 8.94 (2.83)

OUTCOME MEASURES:

1. Primary Outcome: Snoring Severity Scale
Description: The Snoring Severity Scale (SSS) is a 9-point, validated scale to measure the severity of snoring. A total of three questions are asked: 1) "How often do you snore, 2) "How long do you snore", and 3) How audible is your snoring. Answers for each of these questions are summed for a total SSS score. A score of '0' would indicate no snoring at all, while a score of '9' would indicate the most severe snoring as measured by the SSS.
  Outcome measure reported as change with use of the device over pre-trial. In this case, a negative ('-') would represent improvement in snoring symptoms, while a positive ('+') number would indicate an increase in snoring severity.
Time Frame: Baseline and 10 Days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Trial Participants
Number analyzed (Participants) | 570
units on a scale | -4.1 (0.082)
Statistical Analysis 1: Comparison: Clinical Trial Participants; Test type: Superiority; p < 0.0001, t-test, 2 sided — Assuming a priori threshold for statistical significant of p = 0.05

2. Primary Outcome: Visual-Analogue Scale, Self-Reported Snoring Habits
Description: Quantitative assessment on 1-10 scale. Outcome measurement reported as a percentage change from pre-trial with use of the device. A negative ('-') percentage would indicate a reduction in snoring symptoms as measured by the VAS, while a positive percentage ('+') result would indicate an increase in the measured symptom.
Time Frame: Baseline and 10 Days
Measure: Number; unit: percent change
Arm/Group | Clinical Trial Participants
Number analyzed (Participants) | 570
percent change
  How much does your snoring bother YOU? | -51.5
  How much does your snoring bother YOUR PARTNER? | -60.2
  How frequently do you snore? | -56.8
Statistical Analysis 1: Comparison: Clinical Trial Participants; Test type: Superiority; p < 0.0001, t-test, 2 sided — a priori threshold for statistical significance of p = 0.05

ADVERSE EVENTS:
Time Frame: Four months
Arm/Group | Clinical Trial Participants
All-Cause Mortality (participants affected / at risk) | 0/570
Serious Adverse Events (participants affected / at risk) | 0/570
Other Adverse Events (participants affected / at risk) | 1/570
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Trial Participants (N=570)
Device Detached (Product Issues) | 1 (1) — The connection between the top tray and bottom tray was broken, causing the top and bottom trays to detach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03128307/Prot_SAP_000.pdf